CLINICAL TRIAL: NCT07289698
Title: Handgrip Strength Increases the Pressure in the Portal and Left Gastric Veins in Cirrhotic Patients
Status: Recruiting | Type: Observational
Sponsor: Shanxi Provincial People's Hospital (Other Government)
Collaborators: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: MZ
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Handgrip Strength; Transjugular Intrahepatic Portosystemic Shunts (TIPS)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Portal pressure measurement group
  Interventions: Device: Handgrip strength
- Doppler Ultrasound Measurement Group
  Interventions: Device: Handgrip strength

INTERVENTIONS:
Device: Handgrip strength — Jamar Hand Dynamometer, from Illinois, USA. Maximum handgrip strength was measured three times, with each measurement lasting 3 seconds and a 1-minute interval between tests

SUMMARY:
1.Background Handgrip strength , a core indicator of muscle function, has been confirmed to be significantly associated with the clinical prognosis of patients with liver cirrhosis. However, no studies have explored its correlation with portal venous hemodynamics. 2. Objective The purpose of the study is to examine the effects of Handgrip strength on portal vein and left gastric vein pressure, blood flow velocity and direction in patients with liver cirrhosis.

3. Method: observational study. Detection Timing: Doppler ultrasound was employed to determine the portal flow velocity and direction at baseline and during the handgrip strength test in cirrhotic patients with a history of variceal bleeding. Three days later, prior to TIPS placement, the pressures in the portal pressure and gastric vein pressure were measured both before and after handgrip strength. Furthermore, carvedilol and vasoactive drugs were discontinued three days before the study commenced. 4. Elaboration of the Research Hypothesis 4.1. Core Hypothesis The handgrip strength level in patients with liver cirrhosis is correlated with portal venous system hemodynamic indices. Specifically, enhanced handgrip strength may affect portal hypertension and the hemodynamics of varicose veins by improving systemic muscle function or circulatory status. 4.2. Speculation on potential mechanisms Association between muscle function and circulation: As a representative of systemic muscle function, increased handgrip strength may reflect an increase in cardiac output or changes in splanchnic vascular resistance, thereby influencing portal venous hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years of age) with cirrhosis and a history of variceal bleeding, who were preparing for TIPS creation for secondary prophylaxis against variceal bleeding

Exclusion Criteria:

* Severe congestive heart failure, or severe untreated valvular heart disease
* Moderate to severe pulmonary hypertension
* Uncontrolled systemic infection
* Lesions (e.g., cysts) or tumors in the liver parenchyma that preclude TIPS creation
* Overt hepatic encephalopathy
* Unrelieved biliary obstruction
* Child-Pugh score > 13
* Model for end-stage liver disease (MELD) score > 18
* International normalized ratio (INR) > 5
* Platelet count < 20×109/mm3
* Participants who had undergone hand or wrist surgery within the previous 3 months or were unable to hold the dynamometer with the testing hand were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This observational study was performed in two centers in China (The First Affiliated Hospital, and College of Clinical Medicine of Henan University of Science and Technology [Luoyang], and Shanxi Provincial People's Hospital [Taiyuan]) . They serve as the major tertiary referral center for the management of liver cirrhosis and its complications in our country.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
portal pressure | through study completion, an average of 5 minutes
  Prior to TIPS, the pressure monitoring catheter was connected to the pressure-measuring device. Subsequently, the pressures in both the portal vein and left gastric vein were measured simultaneously at baseline and during the handgrip strength test.
left gastric vein pressure | through study completion, an average of 5 minutes
  Prior to TIPS, the pressure monitoring catheter was connected to the pressure-measuring device. Subsequently, the pressures in both the portal vein and left gastric vein were measured simultaneously at baseline and during the handgrip strength test.
portal flow velocity | Before the handgrip strength test, and during the maximum handgrip strength phase, measurements were conducted at intervals of 15 seconds, 30 seconds, 45 seconds, and 60 seconds after the release of strength related to the handgrip Strength
Portal vein blood flow direction | Before the handgrip strength test, and during the maximum handgrip strength phase, measurements were conducted at intervals of 15 seconds, 30 seconds, 45 seconds, and 60 seconds after the release of strength related to the handgrip Strength

SECONDARY OUTCOMES:
Serum albumin (g / l) | Baseline
  Pre-TIPS baseline characteristics ,date (n=32)
alanine aminotransferase(IU / L) | Baseline
  Pre-TIPS baseline characteristics, date (n=32)
aspartate aminotransferase (IU / L) | Baseline
  Pre-TIPS baseline characteristics ,date (n=32)
Total bilirubin (µmol / l) | Baseline
  Pre-TIPS baseline characteristics ,date (n=32)
Prothrombin time (second) | Baseline
  Pre-TIPS baseline characteristics ,date (n=32)
Fasting blood glucose (mmol / l) | Baseline
  Pre-TIPS baseline characteristics ,date (n=32)
triglyceride (mmol / l) | Baseline
  Pre-TIPS baseline characteristics ,date (n=32)
Total cholesterol (mmol / l) | Baseline
  Pre-TIPS baseline characteristics ,date (n=32)
Serum creatinine (µmol / l) | Baseline
  Pre-TIPS baseline characteristics ,date (n=32)
Serum potassium (mmol / l) | Baseline
  Pre-TIPS baseline characteristics ,date (n=32)
Serum sodium (mmol / l) | Baseline
  Pre-TIPS baseline characteristics ,date (n=32)
Serum chloride (mmol / l) | Baseline
  Pre-TIPS baseline characteristics ,date (n=32)
Platelet count (× 109 / mm3) | Baseline
  Pre-TIPS baseline characteristics ,date (n=32)
height | Baseline
weight | Baseline
Model for end-stage liver disease score | Baseline
  Model for end-stage liver disease score: 6-40, the higher scores mean a worse outcome.
Child-Pugh score | Baseline
  Child-Pugh score: 5-15, the higher scores mean a worse outcome
Esophageal varices before endoscopic treatment | Baseline
  The diagnosis of esophageal varices and variceal bleeding in patients is confirmed by upper gastrointestinal endoscopy.
Collateral vessels before TIPS placement | Baseline
  Vascular angiography was performed prior to TIPS placement to diagnose collateral circulation. date (n=32)
Ascites | Baseline
  Prior to TIPS, ascites was evaluated by ultrasound in 32 patients with liver cirrhosis.
Prior overt hepatic encephalopathy | Baseline
Etiology of cirrhosis | Baseline
Age | Baseline
Sex | Baseline

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: Yes
The way of sharing IPD: Sharing and email consultation will begin after December 31, 2027.
  Data collection and Management: Case record forms and electronic data captures.
Supporting Information: Study Protocol
Time Frame: Sharing and email consultation will begin after December 31, 2027